CLINICAL TRIAL: NCT02495987
Title: Adaptations in Subcutaneous and Visceral Adipose Tissue Metabolism During Normal and Pathological Pregnancies
Brief Title: White Adipose Tissue in Pregnancy Study
Acronym: WAT
Status: Active, not recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 14HH2393
Record Dates: First submitted 2015-06-29; First posted 2015-07-14 (Estimated); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: ICP; GDM

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Adipose tissue, serum
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to understand the role of metabolic tissues in the changes of the metabolism of pregnant women and whether this contributes to some women developing metabolic diseases of pregnancy such as gestational diabetes (GDM) or intrahepatic cholestasis of pregnancy (ICP). Samples of adipose tissue will be taken when pregnant women are having caesarean section or laparoscopic procedures.

DETAILED DESCRIPTION:
There is a gradual change in metabolism in pregnancy. This is characterised by a switch from normal levels of cholesterol, glucose and bile acids in early pregnancy to high levels of lipids, glucose and bile acids in late pregnancy. This is important to ensure that nutrients are provided for the growing fetus. However, it results in some women developing metabolic diseases of pregnancy, e.g. gestational diabetes mellitus (GDM) or intrahepatic cholestasis of pregnancy (ICP).

This project aims to understand the role of metabolic tissues in the changes of the metabolism of pregnant women. The investigators are asking for permission to collect samples of adipose tissue (subcutaneous and visceral fat) when women are having surgical procedures. Specifically, the investigators would like to take small samples of fat at two time points:

1. When having a caesarean section (3rd trimester of pregnancy)
2. When having laparoscopic surgery for ectopic pregnancy (1st trimester of pregnancy) Samples will only be taken from women having surgery as part of their clinical care. The investigators are requesting permission to collect samples from women with metabolic diseases of pregnancy (GDM and ICP) and matched controls (women with uncomplicated pregnancy). The investigators will also want to collect blood samples.

There is evidence from non-pregnant individuals (and from animal studies) that the adipose tissue in different parts of the body function in different ways. Subcutaneous fat is typically a fat storage tissue while visceral adipose tissue plays a role in metabolism of fat. The investigators' studies in mice suggest that these different fat stores function differently in pregnancy, and they may play a role in the metabolic changes that cause dyslipidaemia and susceptibility to diabetes mellitus. The investigators aim to identify where there are similar changes in function of adipose tissue in human pregnancy, and whether this contributes to the development of GDM and ICP.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 18-50 years of age
* Uncomplicated pregnancies
* Pathological pregnancies such as Type II Diabetes and ICP

Exclusion Criteria:

* Women treated with immunosuppressive agents, e.g. azathioprine.
* Type 1 diabetes mellitus.
* Long-standing treatment with glucocorticoids, e.g. prednisolone
* Hepatitis C, hepatitis B or HIV.
* Women unable to give consent.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women with or without ICP or GDM
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2015-03; Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
To establish whether there is altered function of subcutaneous and visceral fat in the 1st or 3rd trimester of normal pregnancy, ICP or GDM and whether this is associated with alterations in serum lipids and bile acids | 10 years
  Alterations in subcutaneous and visceral fat messenger RNA (mRNA) will be measured using quantitative PCR by fold-change mRNA expression in reference to the control group: normal pregnancy).

SECONDARY OUTCOMES:
To establish whether there are changes in subcutaneous or visceral fat function associated with altered levels of incretins, free fatty acids or other metabolites of relevance to bile acid, lipid or glucose metabolism. | 10 years
  Altered levels of incretins will be measured by either quantitative PCR looking at mRNA expression of target genes (measured in fold-change mRNA expression in reference to the control group: normal pregnancy), or through metabolite (lipid species) assessment by mass spectrometry, measured in absolute concentration of lipid species per mg fat.
To establish whether there are changes in the histological appearance of subcutaneous or visceral fat in the first or third trimester of normal pregnancy, ICP or GDM | 10 years
  Changes in histological appearance will be assess through hematoxylin and eosin staining. Adipocyte area will be quantified using ImageJ to determine mean, median, range and distribution of adipocytes for each group. Smaller adipocytes typically indicates either reduced lipid uptake, increased lipid export or hyperplasia

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Williamson, MBChB, Principal Investigator — Imperial College London
Locations (2):
- United Kingdom (2):
  - Guy's & St Thomas' NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust Hammersmith, London

IPD SHARING:
Plan to Share IPD: No
We will publish our results and findings in research publications.